CLINICAL TRIAL: NCT03584074
Title: Comparative Study for Decrease of Pain Intensity and Pain Sensitivity Between Pregabalin + COX-2 Inhibitor and COX-2 Inhibitor in Patients With Lumbar Spinal Stenosis: Randomized Controlled Trial
Brief Title: Clinical Trial of Pregabalin and COX2 in Spinal Stenosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Ho-Joong Kim, Associate Professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PreCox2
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2018-07-12 (Actual); Status verified 2018-06

CONDITIONS: Spinal Stenosis Lumbar
Keywords: Pregabalin; Selective COX-2 inhibitor
MeSH Terms: interventions — Pregabalin; Celecoxib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pregabalin and COX-2 inhibitor (Experimental): Pregabalin 75mg BID + Celecoxib 200mg qd
  Interventions: Drug: Pregabalin 75mg; Drug: Celebrex 200Mg Capsule
- COX-2 inhibitor (Active Comparator): Celecoxib 200mg qd
  Interventions: Drug: Celebrex 200Mg Capsule

INTERVENTIONS:
Drug: Pregabalin 75mg — Orally taken twice daily for 8 weeks
  Arms: Pregabalin and COX-2 inhibitor
Drug: Celebrex 200Mg Capsule — Orally taken once daily for 8 weeks

SUMMARY:
Aim of this prospective, single-blind, randomized study was to compare the efficacy of the combination of celecoxib and pregabalin and celecoxib only monotherapy for treatment of chronic low-back pain.

DETAILED DESCRIPTION:
The efficacy and safety of the association of celecoxib [a selective cyclooxygenase-2 (COX-2) inhibitor] and pregabalin (commonly used to control neuropathic pain), compared with monotherapy of each, were evaluated for the treatment of chronic low-back pain, a condition known to be due to neuropathic as well as nociceptive pain mechanisms.

We will compare the efficacy of the combination of a selective COX-2 inhibitor (celecoxib) and an antineuropathic drug, pregabalin, versus celecoxib only monotherapy, in the treatment of spinal stenosis.

Each treatment lasted 8 weeks

Primary outcome is mean pain reduction following different treatments regimes. Secondary outcomes are the changes of pain sensitivity, Oswestry disability index, adverse effects due to the treatments under study.

ELIGIBILITY:
Inclusion Criteria:

* Spinal stenosis

Exclusion Criteria:

* Koval grade >=3
* Other musculoskeletal disorders which cause pain on other joint
* Bleeding risk or ulcer history
* Severe cardiovascular, pulmonary, renal, brain, liver dysfunction

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2019-05-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale | At 8 weeks
  Pain score for low back and lower leg

SECONDARY OUTCOMES:
Pain sensitivity questionnaire (PSQ) | At 8 weeks
  Level of pain sensitivity
Oswestry disability index (ODI) | At 8 weeks
  The self-completed questionnaire contains ten topics concerning intensity of pain, lifting, ability to care for oneself, ability to walk, ability to sit, sexual function, ability to stand, social life, sleep quality, and ability to travel